CLINICAL TRIAL: NCT01097642
Title: Randomized Open-Label Neo-Adjuvant Phase II Study Comparing Ixabepilone (I) Vs. Ixabepilone Plus Cetuximab (IC) in Triple Negative Breast Cancer Patients
Brief Title: Neo-Adjuvant Study in Triple Negative Breast Cancer Patients
Acronym: ICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002243; 0908-0265 (Other: HMRI IRB)
Record Dates: First submitted 2010-03-29; First posted 2010-04-01 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cetuximab; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixabepilone (Active Comparator): Brand name is Ixempra ®; it is an epothilone B analog used in combination with other chemotherapeutics against cancer.
  Interventions: Drug: Ixabepilone
- Ixabepilone plus Cetuximab (Experimental): Cetuximab, brand name Erbitux, is an epidermal growth factor receptor (EGFR) inhibitor and monoclonal antibody used with Ixabepilone against cancer.
  Interventions: Drug: Cetuximab; Drug: Ixabepilone

INTERVENTIONS:
Drug: Cetuximab — Cetuximab will be given at 400mg/m^2 IV over 120 minutes for its initial loading dose on day 1 of the first of four 21 day cycles. It will then be administered on a weekly basis at 250 mg/m^2 IV over 60 minutes.
  Other Names: Erbitux
  Arms: Ixabepilone plus Cetuximab
Drug: Ixabepilone — Ixabepilone will be given at 40mg/m^2 IV over 180 minutes on day 1 of each of four 21 day cycles.
  Other Names: azaepothilone B

SUMMARY:
Ixabepilone and capecitabine combination has demonstrated to be an active regimen in patients with metastatic breast cancer after failing other treatments. Cetuximab is active against tumors expressing epidermal growth factor receptor w/demonstrated activity in head & neck and colorectal tumors and may be effective in some breast cancers known to express EGFR. Study seeks to evaluate Ixabepilone alone or in combination with cetuximab as a an antitumor therapy w/randomization stratified by stage (T1N1-3M0 or T2-4 N0-3M0).

DETAILED DESCRIPTION:
Ixabepilone and capecitabine combination has demonstrated to be an active regimen in patients with metastatic breast cancer (MBC) after failing an anthracycline and a taxane regimen. Cetuximab is active in tumors that express epidermal growth factor receptor (EGFR) with demonstrated activity in head and neck and colorectal tumors. A proportion of breast cancers are known to express EGFR. Cetuximab's mechanism of action suggests the possibility of efficacy in breast cancer patients, and several studies show that it may be efficacious in Triple Negative Breast Cancer (TNBC). This study seeks to evaluate Ixabepilone alone or in combination with cetuximab as a possible way to increase antitumor activity. In this randomized open-label phase II trial, patients will be randomized equally between 1) Ixabepilone or 2) Ixabepilone plus Cetuximab. Randomization will be stratified by disease stage (T1N1-3M0 or T2-4 N0-3M0).

The study's primary objective is to determine the pathologic complete response rate (pCR) (breast and axilla) of Ixabepilone versus Ixabepilone when combined with cetuximab in patients with invasive breast adenocarcinoma T1N1-N3M0 or T2-4 N0-3M0 disease who are triple negative and who are candidates for preoperative chemotherapy. The secondary objectives are to evaluate overall objective response rate in both treatment groups and to assess safety and toxicity of each regimen. There are also tertiary, exploratory objectives that will hopefully allow for the correlation of biomarker expression and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic confirmation of invasive breast carcinoma.
* Patients must have intact primary tumor.
* Patients greater than or equal to 18 years.
* Patients should have T1N1-3M0 or T2-4 N0-3M0.
* Patients with bilateral breast cancer are eligible.
* Patients with second primary breast cancers are eligible.
* Patients should have a Karnofsky performance scale of greater than or equal to 70%.
* Patients must have clinically measurable disease to be treated in the neoadjuvant setting.
* Patients should have adequate bone marrow function, as defined by peripheral granulocyte count of greater than or equal to 1500/mm^3, and platelet count greater than or equal to 100000mm^3.
* Patients must have adequate liver function with a bilirubin within normal laboratory values. Alkaline phosphatase and transaminases (ALT and AST) may be up to 1.5 x upper limit of normal (ULN) of the institution.
* Patients should have adequate renal function with creatinine levels within normal range.
* Patients should have a normal left ventricular ejection fraction (LVEF) of greater than or equal to 50%.
* Negative serum or urine pregnancy test for a woman of childbearing potential (WOCBP).
* WOCBP must use a reliable and appropriate contraceptive method during the study and six months after chemotherapy is completed. WOCBP are women who are not menopausal for 12 months or had no previous surgical sterilization.
* Patients must agree to have study biopsies.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.

Exclusion Criteria:

* Patients with a history of other invasive malignancies diagnosed and treated within the previous 5 years, except non-melanoma skin cancer and non-invasive cervical cancer.
* Her2Neu, ER and PR positive patients should be excluded.
* Patients with Inflammatory breast cancer (IBC) are excluded.
* Patients with an organ allograft or other history of immune compromise.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Chronic treatment with systemic steroids or another immunosuppressive agent.
* A Known history of HIV seropositivity.
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin defined as 1 mg a day).
* Other concurrent and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration).
* Patients with a pre-existing peripheral neuropathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Plan to share data to be determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab
Started | 15 | 25
Completed | 15 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab | Total
Number analyzed (Participants) | 15 | 25 | 40
Age, Continuous [Mean (Full Range); unit: years] | 51 [35 to 68] | 57 [42 to 79] | 55 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 25 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 8 | 18 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 10 | 21 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 25 | 40
Triple Negative Negative Breast Cancer (T1N1-N3M0 or T2-4 N0-3M0) [Count of Participants; unit: Participants] — Staging of Triple Negative Breast Cancer was based on the TNM Staging System (T=tumor size/extent; N=number of nearby lymph nodes that have cancer; M=presence/absence of metastases). Patients were assigned to treatment arms using a stratified blocked randomization, with strata based on disease stage (T1N1-3M0 or T2-4 N0-3M0).
  Participants | 14 | 24 | 38

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The study's primary objective is to determine the pathologic complete response rate (pCR) (breast and axilla) of Ixabepilone versus Ixabepilone when combined with cetuximab in patients with invasive breast adenocarcinoma T1N1-N3M0 or T2-4 N0-3M0 disease who are triple negative and who are candidates for preoperative chemotherapy.
  The criteria used: "Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: one year after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab
Number analyzed (Participants) | 15 | 25
Participants | 2 | 8

2. Secondary Outcome: Recurrence Free Survival (RFS)
Description: The secondary objective is to evaluate the RFS in both treatment groups. The criteria used: "Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: Median 3-year
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab
Number analyzed (Participants) | 15 | 25
Participants | 9 | 17

3. Secondary Outcome: Safety and Toxicity of Both Treatment Regimens: Number of Participants With Adverse Events
Description: The number of participants with adverse events will be measured. Toxicity/safety will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v.3.0). Baseline signs and symptoms will be recorded and followed throughout the trial. Toxicity assessments will be continuous during treatment and the year of follow-up, after which all study drug-related toxicities will be deemed resolved, stabilized, or irreversible. Vital signs will be performed at baseline and will be monitored pre-dose and during study drug administration for Cycles 1 - 4. Chemistry and hematology laboratory tests will be done at baseline and prior to each subsequent chemotherapy cycle.
Time Frame: one year after last treatment dose
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab
Number analyzed (Participants) | 15 | 25
Participants | 15 | 25

ADVERSE EVENTS:
Time Frame: Safety was assessed from time of informed consent signing through 30 days after last treatment dose (an average of 12 weeks).
Arm/Group | Ixabepilone | Ixabepilone Plus Cetuximab
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/15 | 6/25
Other Adverse Events (participants affected / at risk) | 15/15 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=15) | Ixabepilone Plus Cetuximab (N=25)
Peripheral neuropathy (Nervous system disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
GI Events (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=15) | Ixabepilone Plus Cetuximab (N=25)
Anemia (Blood and lymphatic system disorders) | 11 | 18
Fatigue (General disorders) | 10 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT01097642/Prot_SAP_000.pdf